CLINICAL TRIAL: NCT05112952
Title: A Single-Dose, Open-Label, Parallel-Group, Multi-Center Study to Evaluate the Effect of Hepatic Impairment on the Pharmacokinetics of Lazertinib (JNJ-73841937)
Brief Title: A Study to Evaluate the Effect of Hepatic Impairment on Lazertinib (JNJ-73841937)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CR109022; 2021-001950-71 (EudraCT Number); 73841937NSC1007 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2021-11-02; First posted 2021-11-09 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Hepatic Impairment; Healthy
MeSH Terms: interventions — lazertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part A: Group 1: Moderate Hepatic Impairment (Experimental): Participants with moderate hepatic impairment will receive a single oral dose of lazertinib.
  Interventions: Drug: Lazertinib
- Part A: Group 2: Normal Hepatic Function (Active Comparator): Participants with normal hepatic function who qualify for the control group will receive a single oral dose of lazertinib.
  Interventions: Drug: Lazertinib
- Part B: Group 3 (Optional): Mild Hepatic Impairment (Experimental): Participants with mild hepatic impairment will receive a single oral dose of lazertinib.
  Interventions: Drug: Lazertinib
- Part B: Group 4 (Optional): Severe Hepatic Impairment (Experimental): Participants with severe hepatic impairment will receive a single oral dose of lazertinib.
  Interventions: Drug: Lazertinib

INTERVENTIONS:
Drug: Lazertinib — Lazertinib tablet will be administered orally.
  Other Names: JNJ-73841937,; YH25448

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics (PK) of a single oral dose of lazertinib in participants with impaired hepatic function when compared with healthy participants with normal hepatic function, under fed conditions.

ELIGIBILITY:
Inclusion Criteria:

All Participants:

* Must have a clinically stable hepatic function as confirmed by the serum bilirubin and transaminase levels measured during screening and those measured on Day -1
* Willing and able to adhere to the prohibitions and restrictions specified in this protocol
* If a woman, must not be of childbearing potential: postmenopausal (amenorrhea for at least 12 months and a serum follicle stimulating hormone within postmenopausal range); or surgically sterile (hysterectomy, bilateral salpingectomy, bilateral oophorectomy, bilateral tubal occlusion/ligation procedure)

Healthy Participants with normal hepatic function:

* Blood pressure (after the participant is supine for 5 minutes) between 90 and 140 millimeter of mercury (mmHg) systolic for participants less than or equal to (<=) 60 years old and between 90 and 150 mmHg for participants greater than (>) 60 years old, inclusive, and no higher than 90 mmHg diastolic. If blood pressure is out of range, up to 2 repeated assessments are permitted per visit
* Pharmacogenomics: Healthy participants must have matching glutathione S-transferase Mu 1 (GSTM1) genotype (null or non-null GSTM1 genotype) to individual hepatic impairment group participants

Participants with hepatic impairment:

* A 12-lead electrocardiogram (ECG) consistent with adequate cardiac conduction and function as per judgement by the investigator, including: a) Sinus rhythm; b) Heart rate between 50 and 100 beats per minute (extremes included); c) QTc interval <= 480 milliseconds (ms) (corrected cf. Fridericia; QTcF)
* Concomitant medications to treat underlying disease states or medical conditions related to hepatic impairment are allowed. Participants must be on a stable dose of medication and/or treatment regimen for at least 2 weeks before dosing as well as during the study

Exclusion Criteria:

All Participants:

* Participant has known allergies, hypersensitivity, or intolerance to Lazertinib or its excipients
* Any surgical or medical condition that may alter the absorption, metabolism, or excretion of the study drug (example, gastrectomy, Crohn's disease etc.), with the exception of hepatic impairment
* Active gall bladder or biliary tract disease (example, acute cholecystitis, symptomatic cholelithiasis)
* Participant tests positive for human immunodeficiency virus (HIV)-1 or HIV-2 at screening
* Participant has a lack of adequate venous access

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2022-07-11 (Actual); Study Completion 2022-07-11 (Actual)

PRIMARY OUTCOMES:
Plasma Concentrations of Lazertinib | Predose up to 312 hour postdose (up to Day 14)
  Plasma concentrations of lazertinib will be analyzed using a validated, specific, and sensitive method to assess the effect of hepatic impairment on the pharmacokinetic of lazertinib.

SECONDARY OUTCOMES:
Percentage of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | Up to 49 days
  AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non investigational) product. An AE does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (2):
- Germany (2):
  - CRS Clinical Research Services Kiel GmbH, Kiel
  - APEX GmbH, München

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency